CLINICAL TRIAL: NCT01056653
Title: Fathers and Late Preterm Babies Study: Effects of an Educational Intervention on Fathers' Interactions With Infants Born Between 34 and 36 Weeks Gestation
Brief Title: Fathers and Late Preterm Babies Study
Acronym: FLPTB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Karen Benzies, Professor, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: E-21846; ACCFCR Grant # 0802INV-Benzies (Other Grant/Funding Number: Alberta Centre for Child, Family & Community Research)
Record Dates: First submitted 2010-01-22; First posted 2010-01-26 (Estimated); Results first posted 2017-02-23 (Actual); Last update posted 2017-03-29 (Actual); Status verified 2017-02

CONDITIONS: Premature Birth
Keywords: father-child relations; paternal behaviour; early intervention; child-rearing
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group A Teal (Experimental): Standard Dose - Two intervention home visits (at 4 and 6 months of age)
  Interventions: Behavioral: Standard Dose
- Group B Purple (Experimental): High Dose - Four intervention home visits (at 4, 5, 6, and 7 months of age)
  Interventions: Behavioral: High Dose
- Group C Yellow (Sham Comparator): Comparison Group - One home visit, information only (at 4 months of age)
  Interventions: Behavioral: Comparison Group

INTERVENTIONS:
Behavioral: Standard Dose — Two intevention home visits
  Arms: Group A Teal
Behavioral: High Dose — Four intervention home visits
  Arms: Group B Purple
Behavioral: Comparison Group — One home visit, information only
  Arms: Group C Yellow

SUMMARY:
The purpose of this study is to test an educational intervention for first-time fathers of late preterm (34 to 36 weeks gestation) infants.

DETAILED DESCRIPTION:
Background: Preterm birth (PTB) is associated with 75% of morbidity in neonates. Although mortality and morbidity is higher for children with early PTB (< 32 weeks' gestation), late PTB (between 34 to 36 weeks gestation) is more common and creates a serious impact on public health. Indeed, late PTBs constitute 74% of all PTBs, and even modest increases in the rate of late PTB have dramatic effects on health care costs. PTB rates are rising across Canada and in Alberta at an even faster rate: between 1996 and 2005, the rate of PTB in Alberta increased by 23%. Late PTBs accounted for the majority of this increase. While it is clear that early PTB and being small for gestational age (GA) are risk factors for later developmental challenges even into adulthood, the risks and the negative effects of late PTB on child development are emerging. In spite of evidence that heavier weight (and usually older gestation) infants benefit more from early interventions than their lighter weight counterparts, late preterm infants are ineligible for early intervention programs unless they have other health problems. Most programs are designed for mothers, yet fathers contribute to their child's development by providing interactions that are more vigorous, stimulating, and state-disruptive than mothers. Given their increased risk for delays, it is important that both mothers and fathers of late preterm infants are skilled in parent-child interactions to support development. A new intervention for fathers using positive individualized feedback on parent-child interactions has shown promise in improving interactions with healthy infants. However, it is unknown whether this intervention will be effective for fathers of late preterm infants. The purpose of this study is to test an educational intervention for first-time fathers of late preterm (34 to 36 weeks gestation) infants.

Hypothesis: Compared to a comparison group, first-time fathers of late preterm infants who receive an educational intervention will have more positive father-infant interactions when the infant is 8 months old (adjusted age to account for prematurity) as measured during structured play using the Parent Child Interaction Teaching Scale (PCITS) (also known as the Nursing Child Assessment Teaching Scale [NCATS]) scored by raters who are blind to group assignment.

Secondary Research Question: What is the effect of the intervention on fathers' perceptions of parenting stress as measured by the Parenting Stress Index (PSI) at 4 and 8 months adjusted age? Method: In this pilot randomized controlled trial, data will be collected from 148 English speaking, first time fathers of healthy, late preterm, singleton infants. Fathers in the intervention group will receive two home visits when their infant is 4 and 6 months old (adjusted age) and one web-based booster session. Fathers in the comparison group will receive a home visit and discuss a list of age appropriate toys. For all fathers, baseline interactions and parenting stress will be measured at 4 months with outcomes at 8 months.

Measures: The PCITS is an observational measure used to measure changes in father-child interaction after intervention and includes a Parent Domain score composed of sensitivity to cues, response to distress, cognitive growth fostering, and socio-emotional growth fostering. The PSI is a self-report instrument that provides a Parent Domain score reflecting a parent's experience of stress as a parent. The Child Domain score reflects the parental perceptions of the child's temperament and behaviour. All measures have established reliability and validity and inter-rater reliability will be assessed.

Analyses: The socio-demographic and baseline variables will be compared between study groups using descriptive statistics (mean or median when appropriate, standard deviation or interquartile range when appropriate, and proportions). Correlations will be used to determine relationship between the dependent variable (interaction) and any known confounders that may need to be used as covariates. To test our primary hypothesis that differences will exist between groups on father-infant interaction a linear model adjusting for covariates will be used. The same approach will be used to test overall treatment effect on parenting stress in the Parent and Child Domains. We will include subgroup analyses to test for interaction effects between baseline variables and group, and between fathers who did and did not use the web-based booster.

Significance: The results will help in the design of educational interventions to mitigate risks, and optimize developmental outcomes for late preterm infants through enhancing fathers' interactions with their children, and complementing the effects of mothers' contributions to their children's development.

ELIGIBILITY:
Inclusion Criteria:

* Fathers - first-time father, 18 years or older, speak and read English, live with the child's other parent, live within one hours' drive of the university
* Infants - born between 34 weeks and 0 days and 36 weeks and 6 days gestation, singleton

Exclusion Criteria:

* Fathers - known addictions
* Infants - one of a multiple birth, required assisted ventilation, had culture-proven sepsis, major surgical procedure, identified major congenital anomalies, chromosomal anomalies, intracranial hemorrhage, neurologic disorder, or perinatal asphyxia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2008-12; Primary Completion 2012-02 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen M Benzies, PhD, Principal Investigator — University of Calgary
Locations (1):
- University of Calgary, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Benzies K, Magill-Evans J, Harrison MJ, MacPhail S, Kimak C. Strengthening new fathers' skills in interaction with their 5-month-old infants: who benefits from a brief intervention? Public Health Nurs. 2008 Sep-Oct;25(5):431-9. doi: 10.1111/j.1525-1446.2008.00727.x. PMID 18816360
- [Background] Magill-Evans, J., Harrison, M. J., Benzies, K. M., Gierl, M., & Kimak, C. (2007). Effects of parenting education on first-time fathers' skills in interactions with their infants. Fathering, 5, 42-57.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from two Canadian cities between December 2008 and June 2011. There were 1035 fathers that were contacted during birth admission (102 enrolled), from another study (7 enrolled), or from a neonatal database (4 enrolled).
Pre-assignment Details: Potential participants were screened and enlisted at the time of the infant's birth. When the infant was 2.5 months old, additional screening was done and verbal consent secured.
Groups:
- Group A Teal: Two intervention home visits
  Standard Dose: Two home visits (at 4 and 6 months of age)
- Group B Purple: Four home visits
  High Dose: Four home visits (at 4, 5, 6, and 7 months of age)
- Group C Yellow: Comparison Group (information only)
  Comparison Group: One home visit, information only (at 4 months of age)
Period: Overall Study
Arm/Group | Group A Teal | Group B Purple | Group C Yellow
Started | 46 | 23 | 44
Completed | 46 | 23 | 42 (2 were lost to follow-up because one mother left the country and one father was too busy.)
Not Completed | 0 | 0 | 2
Not completed — Lost to Follow-up | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: Sociodemographic and health data were collected with the first home visit.
Groups:
- Group A Teal: Two intervention home visits
  Standard Dose: Two home visits
- Group B Purple: Four home visits
  High Dose: Four home visits
- Group C Yellow: Comparison Group (information only)
  Comparison Group: One home visit, information only
- Total: Total of all reporting groups
Arm/Group | Group A Teal | Group B Purple | Group C Yellow | Total
Number analyzed (Participants) | 46 | 23 | 42 | 111
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.7 (6.44) | 34.28 (4.24) | 34.47 (6.01) | 34.13 (5.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 46 | 23 | 42 | 111
Race/Ethnicity, Customized [Number; unit: participants]
  European | 30 | 19 | 35 | 84
  Filipino | 2 | 0 | 0 | 2
  Chinese | 1 | 0 | 1 | 2
  South Asian | 2 | 2 | 2 | 6
  Arab/West Asian | 1 | 0 | 0 | 1
  Black | 2 | 0 | 1 | 3
  North American First Nations | 2 | 1 | 1 | 4
  Latin American | 1 | 0 | 1 | 2
  Other | 1 | 0 | 1 | 2
  More than one Option Selected | 3 | 0 | 0 | 3
  Did Not Answer | 1 | 1 | 0 | 2
Sex of the Infant [Number; unit: infants]
  Males | 26 | 12 | 25 | 63
  Females | 20 | 11 | 17 | 48
Infants gestational age [Mean (Standard Deviation); unit: days] | 250 (6.27) | 248 (6.40) | 249 (6.61) | 249.08 (6.41)
Education level [Number; unit: participants]
  High school or less | 5 | 2 | 2 | 9
  Partial university/college/technical school | 5 | 4 | 9 | 18
  Completed college/technical school | 12 | 4 | 8 | 24
  University degree | 18 | 8 | 16 | 42
  Postgraduate degree | 6 | 5 | 7 | 18
Household income [Number; unit: participants]
  <$40,000 | 3 | 0 | 2 | 5
  $40,000-$59,999 | 3 | 2 | 3 | 8
  $60,000-$79,999 | 4 | 5 | 0 | 9
  $80,000-$99,999 | 5 | 3 | 6 | 14
  >=$100,000 | 31 | 13 | 31 | 75
Employment Status [Number; unit: participants]
  Working (Full- or part-time) | 44 | 21 | 39 | 104
  On parental leave | 1 | 0 | 1 | 2
  Looking for work | 1 | 1 | 1 | 3
  Going to school | 0 | 0 | 0 | 0
  Caring for family | 0 | 1 | 0 | 1
  Other | 0 | 0 | 1 | 1
Marital Status [Number; unit: participants] — Participants had to be married or living together to be able to participate in the study.
  participants
    Married | 37 | 20 | 35 | 92
    Common law/living with partner/living as married | 9 | 3 | 7 | 19
Main Language Spoken at Home [Number; unit: participants] — Speaking mainly English at home was one of the eligibility criteria. Participants who answered anything but English in the 4 month questionnaire would have indicated at recruitment when their baby was born that they speak mainly English at home.
  participants
    English | 43 | 22 | 40 | 105
    Chinese | 1 | 0 | 0 | 1
    Farsi | 1 | 0 | 0 | 1
    French | 0 | 0 | 1 | 1
    Oriya | 0 | 1 | 0 | 1
    Punjabi | 1 | 0 | 0 | 1
    Spanish | 0 | 0 | 1 | 1
Parent Child Interaction Teaching Scale (PCITS) [Mean (Standard Deviation); unit: Scores on a scale] — Collected when the infant was 4 months old. Assesses parent-infant interaction skills. Used for children from birth to 3 years of age. It is an observational measure of the presence of behaviours in parent-infant interactions.
  The Parent Total (50 items) is the sum of 4 subscales: Sensitivity to Cues (11 items), Response to Distress (11 items), Social-Emotional Growth Fostering (11 items), and Cognitive Growth Fostering (17 items). Higher scores on all subscales and higher total scores reflect more optimal parent-infant interactions.
  Scores on a scale
    Parent Total | 39.72 (4.41) | 40.70 (3.89) | 40.26 (4.13) | 40.13 (4.18)
    Subscale - Sensitivity to Cues | 9.61 (1.37) | 9.52 (1.31) | 9.88 (1.11) | 9.69 (1.26)
    Subscale - Socioemotional Growth Fostering | 8.33 (1.65) | 8.83 (1.30) | 8.69 (1.70) | 8.57 (1.61)
    Subscale - Cognitive Growth Fostering | 11.63 (2.20) | 12.13 (1.91) | 11.52 (2.65) | 11.69 (2.32)
    Subscale - Response to Distress | 10.15 (0.99) | 10.22 (0.80) | 10.17 (0.76) | 10.17 (0.86)
Parenting Stress - Parenting Stress Index - Third Edition (PSI-3) [Mean (Standard Deviation); unit: Scores on a scale] — Collected when the infant was 4 months old.
  A 120-item self-report questionnaire with two domains of parent (51 items) and child (50 items) stress. Higher scores indicate more stress.
  Scores on a scale
    Child Domain | 96.37 (16.78) | 96.57 (17.00) | 96.71 (15.90) | 96.54 (16.35)
    Parent Domain | 107.46 (15.73) | 107.00 (19.73) | 108.60 (19.56) | 107.79 (17.95)
Perceptions of Parenting an Infant - What Being the Parent of a Baby Is Like (WPL-R) Scale [Mean (Standard Deviation); unit: Scores on a scale] — Collected when the infant was 4 months old.
  A 25-item self-report measure that looks at the perceptions the parents have of caring for an infant. There are 3 subscales: Evaluation, Centrality, and Life Change. Each item is on the 9-point scale.
  Higher scores reflect having more of the attribute.
  Scores on a scale
    Evaluation | 7.58 (0.64) | 7.58 (0.72) | 7.52 (0.80) | 7.56 (0.72)
    Centrality | 6.99 (0.81) | 6.47 (0.81) | 6.75 (1.04) | 6.79 (0.92)
    Life Change | 6.77 (1.02) | 6.03 (1.50) | 6.28 (1.39) | 6.43 (1.30)

OUTCOME MEASURES:

1. Primary Outcome: Parent Child Interaction Teaching Scale (PCITS)
Description: Assesses parent-infant interaction skills. Used for children from birth to 3 years of age. It is an observational measure of the presence of behaviours in parent-infant interactions.
  The Parent Total (50 items) is the sum of 4 subscales: Sensitivity to Cues (11 items), Response to Distress (11 items), Social-Emotional Growth Fostering (11 items), and Cognitive Growth Fostering (17 items). Higher scores on all subscales and higher total scores reflect more optimal parent-infant interactions.
  Possible ranges of scores are as follows: Parent Total (0 - 50), Sensitivity to Cues (0 - 11), Response to Distress (0 - 11), Social-Emotional Growth Fostering (0 - 11), and Cognitive Growth Fostering (0 - 17)
Time Frame: When the infant was 8 months old, adjusting for prematurity
Measure: Mean (Standard Deviation); unit: Scores on a scale
Groups:
- Group B Purple: Four intervention home visits
  High Dose: Four home visits
Arm/Group | Group A Teal | Group B Purple | Group C Yellow
Number analyzed (Participants) | 46 | 23 | 42
Scores on a scale
  Parent Total | 40.00 (3.77) | 41.61 (4.03) | 38.83 (4.33)
  Subscale - Sensitivity to Cues | 9.26 (0.98) | 9.17 (0.98) | 9.07 (1.07)
  Subscale - Socioemotional Growth Fostering | 8.07 (1.72) | 9.00 (1.62) | 7.93 (1.44)
  Subscale - Cognitive Growth Fostering | 12.91 (1.98) | 13.52 (2.33) | 12.10 (2.37)
  Subscale - Response to Distress | 9.76 (0.87) | 9.91 (0.95) | 9.74 (0.89)
Statistical Analysis 1: Comparison: Group A Teal vs Group B Purple vs Group C Yellow; ANCOVA - Group Comparison of Parent Total Score on PCITS at 8 months, controlling for scores at baseline (4 months). Group entered as as fixed factor, outcome scores as dependent variable, and baseline scores as covariate; Test type: Superiority or Other; p = 0.03, ANCOVA; F(2,107)=3.48, partial n2=0.061, observed power=0.639
Statistical Analysis 2: Comparison: Group B Purple vs Group C Yellow; Pairwise Group Comparison based on estimated marginal means - Parent Total Scores; Test type: Superiority or Other; p = 0.03, ANOVA — Bonferroni adjustments for multiple comparisons used
Statistical Analysis 3: Comparison: Group A Teal vs Group C Yellow; Pairwise Group Comparison based on estimated marginal means - Parent Total Scores; Test type: Superiority or Other; p = 0.534, ANCOVA — Bonferroni adjustment for multiple comparisons used
Statistical Analysis 4: Comparison: Group A Teal vs Group B Purple vs Group C Yellow; ANCOVA - Group Comparison of Cognitive Growth Fostering Subscale scores at 8 months, controlling for scores at baseline (4 months). Group entered as fixed factor, outcome scores as dependent variable, and baseline scores as covariate; Test type: Superiority or Other; p = 0.047, ANCOVA; F(2,107)=3.145, partial n2=0.056, observed power=0.593
Statistical Analysis 5: Comparison: Group B Purple vs Group C Yellow; Pairwise Group Comparison based on estimated marginal means - Cognitive Growth Fostering Subscale; Test type: Superiority or Other; p = 0.056, ANCOVA — Bonferroni adjustments for multiple comparisons used
Statistical Analysis 6: Comparison: Group A Teal vs Group C Yellow; Pairwise Group Comparison based on estimated marginal means - Cognitive Growth Fostering Subscale; Test type: Superiority or Other; p = 0.267, ANCOVA — Bonferroni adjustments for multiple comparisons used
Statistical Analysis 7: Comparison: Group A Teal vs Group B Purple vs Group C Yellow; ANCOVA - Group Comparison of Socio-Emotional Growth Subscale scores at 8 months, controlling for scores at baseline (4 months). Group entered as fixed factor, outcome scores as dependent variable, and baseline scores as covariate; Test type: Superiority or Other; p = 0.036, ANCOVA; F(2,107)=3.440, partial n2=0.060, observed power=0.634
Statistical Analysis 8: Comparison: Group B Purple vs Group C Yellow; Pairwise Group Comparison based on estimated marginal means - Socio-Emotional Growth Fostering Subscale; Test type: Superiority or Other; p = 0.036, ANCOVA — Bonferroni adjustments for multiple comparisons used
Statistical Analysis 9: Comparison: Group A Teal vs Group C Yellow; Pairwise Group Comparison based on estimated marginal means - Socio-Emotional Growth Fostering Subscale; Test type: Superiority or Other; p = 1.00, ANCOVA — Bonferroni adjustments for multiple comparisons used
Statistical Analysis 10: Comparison: Group A Teal vs Group B Purple vs Group C Yellow; ANCOVA - Group Comparison of Sensitivity to Cues Subscale scores at 8 months, controlling for scores at baseline (4 months). Group entered as fixed factor, outcome scores as dependent variable, and baseline scores as covariate; Test type: Superiority or Other; p = 0.665, ANCOVA; F(2,107)=0.409
Statistical Analysis 11: Comparison: Group A Teal vs Group B Purple vs Group C Yellow; ANCOVA - Group Comparison of Response to Distress Subscale scores at 8 months, controlling for scores at baseline (4 months). Group entered as fixed factor, outcome scores as dependent variable, and baseline scores as covariate; Test type: Superiority or Other; p = 0.732, ANCOVA; F(2,107)=0.313

2. Secondary Outcome: Parenting Stress - Parenting Stress Index - Third Edition (PSI-3)
Description: A 120-item self-report questionnaire of parenting stress with two domains. The Parent Domain (51 items) measures stress related to parental functioning, the Child Domain (50 items) measures child qualities and characteristics that contribute to stress in the parent-child system. The PSI-3 contains an additional Life Stress scale (19 items) which was not used in the study.
  The range of possible scores in the Parent Domain is 50 - 250 and in the Child Domain is 51 - 255. In both domains, higher scores indicate more stress.
Time Frame: When the infant was 8 months old, adjusting for prematurity
Population: Group A Teal n = 44 due to missing data
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Group A Teal | Group B Purple | Group C Yellow
Number analyzed (Participants) | 44 | 23 | 42
Scores on a scale
  Child Domain | 93.52 (14.83) | 89.96 (16.65) | 93.26 (13.43)
  Parent Domain | 106.48 (15.51) | 103.52 (18.37) | 107.12 (20.46)
Statistical Analysis 1: Comparison: Group A Teal vs Group B Purple vs Group C Yellow; ANCOVA - Group Comparison of Parent Domain scores at 8 months, controlling for scores at baseline (4 months). Group entered as fixed factor, outcome scores as dependent variable, and baseline scores as covariate; Test type: Superiority or Other; p = 0.61, ANCOVA; F(2,107)=0.49
Statistical Analysis 2: Comparison: Group A Teal vs Group B Purple vs Group C Yellow; ANCOVA - Group Comparison of Child Domain scores at 8 months, controlling for scores at baseline (4 months). Group entered as fixed factor, outcome scores as dependent variable, and baseline scores as covariate; Test type: Superiority or Other; p = 0.38, ANCOVA; F(2,107)=0.96

3. Secondary Outcome: Perceptions of Parenting an Infant - What Being the Parent of a Baby Is Like (WPL-R) Scale
Description: 25-item self-report measure composed of 3 subscales: Evaluation (11 items), Centrality (8 items), and Life Change (6 items). Each item is rated on a 9-point scale and subscale scores are obtained by averaging the scores of all items on a subscale; the range for all subscales is therefore 1 - 9. Higher scores reflect having more of the attribute being measured.
Time Frame: When the infant was 8 months old, adjusting for prematurity
Population: Goup A Teal n = 45 due to missing data
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Group A Teal | Group B Purple | Group C Yellow
Number analyzed (Participants) | 45 | 23 | 42
Scores on a scale
  Evaluation | 7.77 (0.54) | 7.97 (0.48) | 7.85 (0.52)
  Centrality | 6.85 (0.84) | 6.48 (1.04) | 6.58 (0.79)
  Life Change | 6.74 (1.12) | 5.93 (1.41) | 6.58 (1.14)
Statistical Analysis 1: Comparison: Group A Teal vs Group B Purple vs Group C Yellow; ANCOVA - Group Comparison of WPL-R scores - Evaluation Subscale scores at 8 months, controlling for scores at baseline (4 months). Group entered as fixed factor, outcome scores as dependent variable, and baseline scores as covariate; Test type: Superiority or Other; p = 0.11, ANCOVA; F(2,106)=2.24
Statistical Analysis 2: Comparison: Group A Teal vs Group B Purple vs Group C Yellow; ANCOVA - Group Comparison of WPL-R scores - Centrality Subscale scores at 8 months, controlling for scores at baseline (4 months). Group entered as fixed factor, outcome scores as dependent variable, and baseline scores as covariate; Test type: Superiority or Other; p = 0.686, ANCOVA; F(2,106)=0.379
Statistical Analysis 3: Comparison: Group A Teal vs Group B Purple vs Group C Yellow; ANCOVA - Group Comparison of WPL-R scores - Life Change Subscale scores at 8 months, controlling for scores at baseline (4 months). Group entered as fixed factor, outcome scores as dependent variable, and baseline scores as covariate; Test type: Superiority or Other; p = 0.121, ANCOVA; F(2,106)=2.158

ADVERSE EVENTS:
Arm/Group | Group A Teal | Group B Purple | Group C Yellow
Serious Adverse Events (participants affected / at risk) | 0/46 | 0/23 | 0/42
Other Adverse Events (participants affected / at risk) | 0/46 | 0/23 | 0/42

LIMITATIONS AND CAVEATS:
Challenges recruiting first-time fathers of late preterm infants; recruiting challenges led to a smaller sample than planned.

Limited inter-rater reliability.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No